CLINICAL TRIAL: NCT03276910
Title: Evaluation of Erythroferrone as a New Biomarker of Erythropoesis Stimulating Agents
Acronym: ERYTHROFER-01
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Association Athletes For Transparency (Other)
Collaborators: University of Milan School of Medicine (Unknown); Centre d'Investigation Clinique Lyon (CIC) (Unknown); Ecole Nationale de Ski et d'Alpinisme (ENSA) (Unknown); Partnership for Clean Competition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Athletes For Transparency
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Sports Drug Abuse
Keywords: antidoping
MeSH Terms: interventions — Epoetin Alfa

STUDY DESIGN:
Intervention Model Description: 3 different conditions:
  * Eprex 20 UI/kg
  * Eprex 50 UI/kg
  * Placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eprex 20 UI/kg (Experimental): 6 doses at 20 IU/kg in subcutaneous use
  Interventions: Drug: EPREX
- Eprex 50 UI/kg (Experimental): 6 doses at 50 IU/kg in subcutaneous use
  Interventions: Drug: EPREX
- Placebo (Placebo Comparator): 6 injections at 1ml in subcutaneous use of sodium chloride AGUETTANT 0.9%
  Interventions: Drug: sodium chloride AGUETTANT 0.9%

INTERVENTIONS:
Drug: EPREX — 6 doses at 50 IU/kg or 20 IU/kg in subcutaneous use
  Arms: Eprex 20 UI/kg; Eprex 50 UI/kg
Drug: sodium chloride AGUETTANT 0.9% — 6 injections at 1ml in subcutaneous use
  Arms: Placebo

SUMMARY:
The main objective of this research is to demonstrate the possible use of erythroferrone (ERFE) as a potential marker of recombinant human erythropoietin (rHuEpo) use to be included in the Athlete Biological Passport (PBA) developed by the World Anti-Doping Agency (WADA).

ELIGIBILITY:
Inclusion Criteria:

* Man between 18 and 49 years old
* Beneficiary of a social protection scheme
* Able to sign informed consent

Exclusion Criteria:

* Hematocrite>50% or Hemoglobin> 17d/dl or Ferritin<30 ug/l
* Hypersensitivity to the active substance or to any of the excipients ofEPREX
* Erythroblastopenia already reported following treatment with erythropoietin
* Uncontrolled hypertension
* Any medication taken as part of a chronic treatment
* Absence of stable or evolutionary pathology without treatment
* History of convulsion or epilepsy
* History of thrombotic vascular events
* Large blood loss due to an accident, pathological condition or other similar situation.
* Donation of blood or blood transfusion within three months prior to inclusion in the protocol.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-09-08 (Estimated); Primary Completion 2017-12-22 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Erythroferrone | 12 measures in 29 days
  dosage Erythroferrone from blood samples

SECONDARY OUTCOMES:
Hbmass | 2 measures in 29 days
  Measure of the total mass of hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Catherine MD CORNU, phD, Principal Investigator — Centre d'Investigation Clinique (CIC)

IPD SHARING:
Plan to Share IPD: Undecided